CLINICAL TRIAL: NCT04176770
Title: ESP Versus TAP for Analgesia After Laparoscopic Cholecystectomy
Brief Title: Comparaison of ESP Block and TAP Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, professor, head of the anesthesia and ICU departement, Mongi Slim Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESP in cholecystectomy
Record Dates: First submitted 2019-11-22; First posted 2019-11-25 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Post Operative Pain
Keywords: Laparoscopic cholecystectomy; Post Operative; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP group (Experimental): ESP block: bilateral injection of 20 ml of isobaric Bupivacain 0,375% in the paraverebral space T5.
  Interventions: Procedure: ESP Block
- TAP Block (Experimental): TAP block: bilateral injection of 15 ml of Isobaric Bupivacain 0,5%
  Interventions: Procedure: TAP Block

INTERVENTIONS:
Procedure: ESP Block — ESP block: bilateral injection of 20 ml of isobaric Bupivacain 0,375% in the paraverebral space T5.
  Arms: ESP group
Procedure: TAP Block — TAP block: bilateral injection of 15 ml of Isobaric Bupivacain 0,5%
  Arms: TAP Block

SUMMARY:
This study aim to compare the efficiency and the analgesic effect of Erector Spinal Plane Block versus TAP Block after laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
This study will include patients scheduled for laparoscopic cholecystectomy, ASA status 1 or 2. patients will be randomized in 2 groups to recieve post operative analgesia with -ESP block: bilateral injection of 20 ml of isobaric Bupivacain 0,375% in the paraverebral space T5.

or

-TAP block: bilateral injection of 15 ml of Isobaric Bupivacain 0,5%

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* ASA status I or II
* scheduled for laparoscopic cholecystectomy

Exclusion Criteria:

* laparotomy
* unplanned ICU admission

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Post Operative analgesia | 24 hours after intervention
  Post operative analgesia assessed with Numerical rating scale (0=minimum, 10= Maximum)

SECONDARY OUTCOMES:
post operative analgesic consumption | 24 hours after intervention
  Amount of Morphin needed for analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Mhamed Sami Mebazaa, Professor, Principal Investigator — Mongi Slim Hospital
Locations (1):
- Mongi Slim Hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No